CLINICAL TRIAL: NCT01751087
Title: Cervical Preparation Before Dilation and Evacuation in the Second Trimester: A Multicenter Randomized Trial Comparing Osmotic Dilators Alone to Dilators Plus Adjunctive Misoprostol or Adjunctive Mifepristone.
Brief Title: Cervical Preparation Before Dilation and Evacuation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood League of Massachusetts (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9-500-25.1; SFPRF6-MS (Other Grant/Funding Number: Society for Family Planning Research Fund); NCT01799928 (obsolete NCT alias)
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Abortion, Induced
Keywords: abortion, induced
MeSH Terms: interventions — Mifepristone; Misoprostol; Ascorbic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Osmotic dilators + placebo (vit c) + placebo (vit B12) (Other): Women will receive osmotic dilators on Day 1, oral placebo on Day 1, and buccal placebo on Day 2.
  Interventions: Device: Osmotic dilators; Other: placebo
- Osmotic dilators + placebo (vit c) + misoprostol (Active Comparator): Women will receive osmotic dilators on Day 1, oral placebo on Day 1, and buccal misoprostol 400 mcg on Day 2.
  Interventions: Drug: misoprostol; Device: Osmotic dilators; Other: placebo
- Osmotic dilators + mifepristone + placebo (vit B12) (Active Comparator): Women will receive osmotic dilators on Day 1, oral mifepristone 200 mg on Day 1, and buccal placebo on Day 2.
  Interventions: Other: Mifepristone; Device: Osmotic dilators; Other: placebo

INTERVENTIONS:
Other: Mifepristone — oral mifepristone 200 mg on Day 1.
  Other Names: Mifeprex
  Arms: Osmotic dilators + mifepristone + placebo (vit B12)
Drug: misoprostol — buccal misoprostol 400 mcg on Day 2
  Other Names: Cytotec
  Arms: Osmotic dilators + placebo (vit c) + misoprostol
Device: Osmotic dilators — osmotic dilators on Day 1
  Other Names: laminaria; Dilapan-S
Other: placebo — placebo for mifepristone, on day 1
  Other Names: vitamin C 500 mg
  Arms: Osmotic dilators + placebo (vit c) + misoprostol; Osmotic dilators + placebo (vit c) + placebo (vit B12)
Other: placebo — placebo for misoprostol, on day 2
  Other Names: vitamin B12 500 mcg
  Arms: Osmotic dilators + mifepristone + placebo (vit B12); Osmotic dilators + placebo (vit c) + placebo (vit B12)

SUMMARY:
The purpose of this research study is to compare three different ways of opening a woman's cervix before her second-trimester surgical abortion.

* Osmotic dilators: small rods that, when inserted into the cervix, gently expand to open the cervix
* Osmotic dilators plus mifepristone, a medicine that is swallowed
* Osmotic dilators plus misoprostol, a medicine that is placed between the cheek and gum

Hypotheses:

* adding buccal misoprostol 3 hours preoperatively will significantly improve dilation compared to laminaria alone, making procedures faster, easier and safer.
* adding oral mifepristone at the time of laminaria placement will confer a similar benefit.
* the efficacy of adjunctive misoprostol and mifepristone will be influenced by gestational age, with women later in gestation having increased efficacy from these agents.
* significantly more patients who receive adjunctive misoprostol or mifepristone will have adequate initial dilation, fewer will require manual dilation or additional cervical preparation and there will be fewer complications in these arms, although complication rates will be low and we will only be able to detect relatively large differences.
* patients will prefer to have the procedure done as quickly as possible with as little discomfort as possible, that cervical ripening with adjunctive misoprostol will be associated with more cramping than osmotic dilators alone and that mifepristone will be well tolerated and may not cause more cramping or other side effects than osmotic dilators alone.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Able to give informed consent
* Medically eligible for outpatient second trimester pregnancy termination at the clinical site
* English-speaking or Spanish-speaking at sites with ability to obtain informed consent in Spanish

Exclusion Criteria:

* Active bleeding (>1 pad/hour) or hemodynamically unstable at enrollment
* Signs of chorioamnionitis or clinical infection at enrollment
* Signs of spontaneous labor or cervical insufficiency at enrollment
* Spontaneous intrauterine fetal demise
* Patient incarcerated
* Allergy to mifepristone or misoprostol
* Chronic steroid use or adrenal insufficiency
* Porphyria
* Inflammatory bowel disease requiring treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, MPH, Principal Investigator — Planned Parenthood League of Massachusetts
Locations (7):
- United States (7):
  - San Francisco General Hospital, San Francisco, California
  - Family Planning Associates, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Planned Parenthood of New York City, New York, New York
  - Lovejoy Surgical Center, Portland, Oregon
  - Magee Women's Hospital, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Goldberg AB, Fortin JA, Drey EA, Dean G, Lichtenberg ES, Bednarek PH, Chen BA, Dutton C, McKetta S, Maurer R, Winikoff B, Fitzmaurice GM. Cervical Preparation Before Dilation and Evacuation Using Adjunctive Misoprostol or Mifepristone Compared With Overnight Osmotic Dilators Alone: A Randomized Controlled Trial. Obstet Gynecol. 2015 Sep;126(3):599-609. doi: 10.1097/AOG.0000000000000977. PMID 26196084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: February 2013-February 2014
  Number of recruitment sites: 7
  Types of location: medical clinic (3), hospital-based (4)
Period: Overall Study
Arm/Group | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) | Osmotic Dilators + Placebo (Vit c) + Misoprostol | Osmotic Dilators + Mifepristone + Placebo (Vit B12)
Started | 100 | 100 | 100
Completed | 99 | 100 | 99
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) | Osmotic Dilators + Placebo (Vit c) + Misoprostol | Osmotic Dilators + Mifepristone + Placebo (Vit B12) | Total
Number analyzed (Participants) | 100 | 100 | 100 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (5.7) | 25.9 (5.9) | 25.3 (5.8) | 25.25 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 100 | 300
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latina | 19 | 18 | 22 | 59
  African American or black | 39 | 48 | 36 | 123
  White or European American | 31 | 22 | 29 | 82
  Other | 11 | 12 | 13 | 36
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 100 | 300

OUTCOME MEASURES:

1. Primary Outcome: Operative Time
Description: The duration of the D&E procedure was measured with a stopwatch, starting with the first instrument that passes into the uterus and ending when the last instrument is removed from the uterus upon completion of the D&E
Time Frame: participants were assessed for the duration of the procedure, an average of 6 minutes
Population: Arm 1 (dilators-alone): 1 subject excluded [withdrawn/no intervention]. Arm 2 (dilators + misoprostol): 2 excluded: [one expelled, no D&E, one D&E not completed on first attempt & data missing]. Arm 3 (dilators + mifepristone): 2 excluded (1 withdrawn/no intervention, 1 D&E not completed on first attempt & data missing].
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) | Osmotic Dilators + Placebo (Vit c) + Misoprostol | Osmotic Dilators + Mifepristone + Placebo (Vit B12)
Number analyzed (Participants) | 99 | 98 | 98
minutes | 6.27 (3.5) | 6.28 (4.6) | 5.53 (2.9)

2. Secondary Outcome: Initial Cervical Dilation
Description: Measured at the time of procedure (immediately before the start of D&E)
Time Frame: participants were assessed during cervical dilation process, average time of 1 minute
Population: Arm 1: 1 subject excluded [withdrawn/no intervention]. Arm 2: 2 excluded: [one expelled, no D&E, one D&E not completed on first attempt & data missing]. Arm 3: 2 excluded (1 withdrawn/no intervention, 1 D&E not completed on first attempt & data missing]. Additionally missing data for one more subject in Arm 2.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) | Osmotic Dilators + Placebo (Vit c) + Misoprostol | Osmotic Dilators + Mifepristone + Placebo (Vit B12)
Number analyzed (Participants) | 99 | 97 | 98
centimeters | 2.2 (0.5) | 2.5 (0.9) | 2.4 (0.5)

3. Secondary Outcome: Ability to Complete the D&E on the First Attempt
Description: Assessed on day of procedure and following day. If the procedure was unable to be completed as planned and the subject had to leave the procedure room and return for another attempt either at a time later the same day or the next day.
Time Frame: participants were assessed for the duration of the procedure, an average of 6 minutes
Measure: Number; unit: participants
Arm/Group | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) | Osmotic Dilators + Placebo (Vit c) + Misoprostol | Osmotic Dilators + Mifepristone + Placebo (Vit B12)
Number analyzed (Participants) | 99 | 100 | 99
participants | 98 | 98 | 98

4. Secondary Outcome: Need for Mechanical Dilation
Description: Assessed on Day of procedure. Assessed immediately after completion of D&E
Time Frame: participants were assessed for the duration of the procedure, an average of 6 minutes
Population: Arm 1: one subject withdrawn/no intervention. Arm 2: one subject expelled, no D&E. Arm 3: one subject withdrawn/no intervention
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) | Osmotic Dilators + Placebo (Vit c) + Misoprostol | Osmotic Dilators + Mifepristone + Placebo (Vit B12)
Number analyzed (Participants) | 98 | 99 | 99
participants | 26 [17.8 to 35.3] | 9 [3.4 to 14.8] | 16 [8.9 to 23.4]

5. Secondary Outcome: Ease of Mechanical Dilation
Description: Number of participants for whom, if additional mechanical dilation was required, it was difficult or very difficult. Assessed on day of procedure. Assessed after completion of D&E
Time Frame: participants were assessed for the duration of the procedure, an average of 6 minutes
Population: Number of participants in each arm who required additional mechanical dilation
Measure: Number; unit: participants
Arm/Group | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) | Osmotic Dilators + Placebo (Vit c) + Misoprostol | Osmotic Dilators + Mifepristone + Placebo (Vit B12)
Number analyzed (Participants) | 26 | 9 | 16
participants | 6 | 4 | 1

6. Secondary Outcome: Complications From Procedure
Description: Patient having any complication, including hospitalizations transfusions additional unplanned procedures
Time Frame: assessed immediately after completion of D&E and at 1 week and 1 month post-procedure
Measure: Number; unit: participants
Arm/Group | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) | Osmotic Dilators + Placebo (Vit c) + Misoprostol | Osmotic Dilators + Mifepristone + Placebo (Vit B12)
Number analyzed (Participants) | 99 | 100 | 99
participants | 10 | 2 | 2

7. Secondary Outcome: Chills (Any) After Day 2 Medication Administration
Description: chills (any) after Day 2 medication administration
Time Frame: assessed immediately after administration of day 2 medication
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) | Osmotic Dilators + Placebo (Vit c) + Misoprostol | Osmotic Dilators + Mifepristone + Placebo (Vit B12)
Number analyzed (Participants) | 99 | 100 | 99
participants | 12 [5.7 to 18.6] | 39 [29.4 to 48.6] | 18 [10.6 to 25.8]

8. Secondary Outcome: Patient Satisfaction With Cervical Prep
Description: Patients who were very satisfied or satisfied with cervical preparation. Assessed on Day of procedure. Assessed after completion of D&E procedure and just prior to discharge home.
Time Frame: patients' satisfaction with cervical prep was evaluated over course of cervical prep and procedure, up to 3 days
Measure: Number; unit: participants
Arm/Group | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) | Osmotic Dilators + Placebo (Vit c) + Misoprostol | Osmotic Dilators + Mifepristone + Placebo (Vit B12)
Number analyzed (Participants) | 99 | 100 | 99
participants | 72 | 80 | 80

9. Secondary Outcome: Physician Satisfaction With Cervical Preparation
Description: Participants for whom the operating physician reported being satisfied or very satisfied with the cervical preparation. Assessed on Day of procedure. Assessed after completion of D&E procedure.
Time Frame: physicians' satisfaction with cervical prep was evaluated over course of procedure, an average of 6 minutes
Population: Data on whether the physician was satisfied with the cervical preparation is available for all participants except:
  Arm 1: 1 participant withdrawn with no intervention; Arm 2: 1 participant who didn't have a D&E (expelled), Arm 3: 1 participant withdrawn with no intervention and one with missing data.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) | Osmotic Dilators + Placebo (Vit c) + Misoprostol | Osmotic Dilators + Mifepristone + Placebo (Vit B12)
Number analyzed (Participants) | 99 | 99 | 98
participants | 71 [62.9 to 80.6] | 78 [70.7 to 86.8] | 85 [80.0 to 93.5]

ADVERSE EVENTS:
Time Frame: 1 month post-procedure
Arm/Group | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) | Osmotic Dilators + Placebo (Vit c) + Misoprostol | Osmotic Dilators + Mifepristone + Placebo (Vit B12)
Serious Adverse Events (participants affected / at risk) | 2/99 | 1/100 | 1/99
Other Adverse Events (participants affected / at risk) | 8/99 | 1/100 | 1/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) (N=99) | Osmotic Dilators + Placebo (Vit c) + Misoprostol (N=100) | Osmotic Dilators + Mifepristone + Placebo (Vit B12) (N=99)
Hospitalization for bleeding (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1)
Hospitalization for bleeding + Hysterectomy (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osmotic Dilators + Placebo (Vit c) + Placebo (Vit B12) (N=99) | Osmotic Dilators + Placebo (Vit c) + Misoprostol (N=100) | Osmotic Dilators + Mifepristone + Placebo (Vit B12) (N=99)
uterine re-aspiration (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 1 (1)
Intrauterine tamponade or cervical stay sutures (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0)
cervical laceration requiring sutures (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations include inadequate sample size to measure complications as a primary outcome and reliance on outcomes that measure efficacy of the cervical preparation rather than its direct effect on overall safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No